CLINICAL TRIAL: NCT00416247
Title: Effect of Hypnosis on Motor Cortex Excitability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Ehud Klein, MD, Head Department of Psychiatry, Rambam Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rambam2409_CTIL
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2006-12

CONDITIONS: Healthy
Keywords: Hypnosis; TMS; Cortical excitability
MeSH Terms: interventions — Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — Hypnosis

SUMMARY:
This study is intended to investigate neurophysiological mechanisms of hypnosis using transcranial magnetic stimulation (TMS) and assessment of motor cortex excitability in healthy volunteers under hypnosis.

ELIGIBILITY:
Inclusion Criteria: .

1. Healthy volunteers aged 20 to 45 years.
2. Hypnotisability above 14 as measured by the Tellegan absorption scale.

Exclusion Criteria:

1. Psychiatric diagnosis in axis I or axis II;
2. Documented history of head injury or seizure disorder;
3. Evidence of a disorder which could affect peripheral and central conduction such as multiple sclerosis, motor neuron disease, carpal tunnel syndrome, cervical spondylosis, diabetic neuropathy.
4. Any other contraindication to TMS as specified in the safety guidelines for rTMS (Wassermann, 1998) such as cardiac pacemakers or metallic deep brain electrodes.
5. Chronic pharmacological treatment.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cortical Excitability | Before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Klein, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel